CLINICAL TRIAL: NCT07008430
Title: Angle-Specific Torque Profiles of Wrist, Forearm and Elbow Movements After Distal Radius Fracture
Brief Title: Angle Specific Torque Profiles After Distal Radius Fracture
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Barış SEVEN, Ph.D, Izmir Katip Celebi University
Other Study IDs: 8
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Radius Distal Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — There will be no intervention. Only archival data will be analyzed

SUMMARY:
Distal radius fracture (DRF) is one of the most common upper extremity injuries and can lead to long-term kinesiological and anatomical alterations despite proper surgical fixation and rehabilitation. This retrospective cohort study aims to analyze the angle-specific torque characteristics of wrist (flexion/extension), forearm (supination/pronation), and elbow (flexion/extension) movements in patients with a history of DRF treated by volar plate fixation.

The study will utilize archived raw data of 37 eligible patients who underwent isokinetic strength testing during the post-rehabilitation period. Data will be extracted from Cybex NORM® and Humac isokinetic dynamometer systems and analyzed using Statistical Parametric Mapping (SPM) with the open-source spm1d package in MATLAB. This analysis will generate 101-point angle-dependent torque curves for each joint movement and will be used to evaluate interlimb asymmetry, angle of peak torque production, and unilateral agonist/antagonist torque ratios.

Additionally, radiographic images archived during the treatment period will be analyzed to measure radial inclination, palmar tilt, and ulnar variance using the Dresdner scoring system. The torque profiles and radiological parameters will be statistically analyzed with SPSS. Between-limb comparisons and symmetry indices will be calculated using repeated-measures ANOVA, t-tests or non-parametric alternatives, depending on data distribution.

This research is expected to provide new insights into the kinesiological consequences of DRF by presenting detailed angle-specific torque characteristics, going beyond conventional peak torque and range of motion assessments commonly seen in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal radius fractures reduced with a volar plate will be included.

Exclusion Criteria:

* Patients with bilateral injuries, fractures in bones other than the radius, stabilization methods other than volar plate, and any other neurological or orthopedic condition that may affect the evaluation will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with distal radius fracture
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Angle Specific Torque Profiles | 1 year
  Raw data files of both the injured and uninjured upper limbs of eligible patients will be obtained from the system records of the isokinetic dynamometer. These raw data will be analyzed using the open-source spm1d package within the MATLAB software (R2021b, The MathWorks Inc., Natick, MA) through statistical parametric mapping (SPM). Accordingly, torque/angle data produced during the full range of motion on the isokinetic dynamometer will be divided into 101 intervals to construct angle-dependent torque profiles (SPM analysis) for each movement.
  SPM analysis will be conducted for wrist flexors and extensors, forearm supinators and pronators, and elbow flexors and extensors. Through this analysis, the following parameters will be examined: the angle-dependent torque characteristics of the injured and uninjured limbs, the unilateral angle-dependent agonist/antagonist torque profiles, and the angle at which peak torque occurs.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided